CLINICAL TRIAL: NCT04372173
Title: A Comprehensive Evaluation of Thrombotic/Fibrinolytic Activation Before and After Total Hip Arthroplasty
Brief Title: An Evaluation of Clotting Factor Activity Before and After Total Hip Arthroplasty
Acronym: CloFaTHA
Status: Completed | Type: Observational
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Dariusz Tomaszewski, MD, PhD, Adjunct Professor, Military Institute od Medicine National Research Institute
Other Study IDs: 681006-7
Record Dates: First submitted 2020-04-14; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Arthroplasty, Replacement; Coagulation Factors
Keywords: total hip arthroplasty; coagulation factors; venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: analysis of the concentration of the clotting factors in patients who underwent primary hip arthroplasty — Blood samples were taken before surgery, 6 hours, two, four, and six days after the procedure. Venous blood samples were taken from peripheral veins.
  All analyzed parameters (fibrinogen, factor II, factor VIII, factor X, D-dimer) were determined using an ACL TOP 500 CTS automated coagulation analyzer.
  All patients were operated on by a single surgical team, with cementless hip replacements implanted, and without tranexamic acid administered in the perioperative period. All patients underwent venous thromboembolic complications prophylaxis.
  The following data were collected: age, body mass index, gender, perioperative risk assessment scale according to the American Society of Anesthesiologists score, blood transfusions, hemoglobin levels before surgery and two days post-surgery, instances of thromboembolic complications. Because of the observational nature of this study no changes in the treatment of patients were made.

SUMMARY:
The objective of the study was to analyze both the concentration and the activity of the clotting factors, D-dimer levels, as well as fibrinogen concentration in patients who underwent primary total hip arthroplasty due to idiopathic arthrosis.

Blood loss is often related to perioperative period and may result in decrease of concentration of coagulation factors, which in turn may lead to increased bleeding. We analyzed data of thirty patients scheduled for primary hip arthroplasty: the activity of clotting factors II, VIII, X, as well as fibrinogen concentration in the following time points: (i) before surgery, (ii) six hours after the procedure, and (iii) two, (iv) four, and (v) six days after the operation. All laboratory tests were performed using automatic analyzer. At the same time intervals, an immunoenzymatic assay was used to determine D-dimer levels.

ELIGIBILITY:
Inclusion Criteria:

* patients qualified for primary hip arthroplasty for idiopathic osteoarthritis

Exclusion Criteria:

* hip osteoarthritis because of non-idiopathic etiology
* history of venous thromboembolism or arterial embolism
* anticoagulation treatment,
* coagulopathy
* infection, and
* renal failure defined as a creatinine clearance below 50 ml/minute.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There were 12 men and 18 women in the study group. Mean age: 67 years. Mean body mass index: 26. Mean ASA score: II.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Changes of serum fibrinogen | This measure will be measured (1) before surgery, (2) six hours after the procedure; (3) second, (4) fourth, and (5) sixth day after the operation
  Serum fibrinogen concentration will be measured (1) before surgery, (2) six hours after the procedure; (3) second, (4) fourth, and (5) sixth day after the operation
Changes of coagulation factor II | This measure will be measured (1) before surgery, (2) six hours after the procedure; (3) second, (4) fourth, and (5) sixth day after the operation
  Activity of the coagulation factor II will be measured (1) before surgery, (2) six hours after the procedure; (3) second, (4) fourth, and (5) sixth day after the operation
Changes of coagulation factor VIII | This measure will be measured (1) before surgery, (2) six hours after the procedure; (3) second, (4) fourth, and (5) sixth day after the operationixth day after the operation
  Activity of the coagulation factor VIII will be measured (1) before surgery, (2) six hours after the procedure; (3) second, (4) fourth, and (5) sixth day after the operation
Changes of coagulation factor X | This measure will be measured (1) before surgery, (2) six hours after the procedure; (3) second, (4) fourth, and (5) sixth day after the operation
  Activity of the coagulation factor X will be measured (1) before surgery, (2) six hours after the procedure; (3) second, (4) fourth, and (5) sixth day after the operation
Changes of D-dimer | This measure will be measured (1) before surgery, (2) six hours after the procedure; (3) second, (4) fourth, and (5) sixth day after the operation
  Blood concentration of the D-dimer will be measured (1) before surgery, (2) six hours after the procedure; (3) second, (4) fourth, and (5) sixth day after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Therapy, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided